CLINICAL TRIAL: NCT06802900
Title: Assessment of Surgical Techniques and Clinical Outcomes in Patients Undergoing Nerve-Sparing Modified Radical Hysterectomy with Uterine Skeletonization for Deep Infiltrative Endometriosis (DIE)"
Brief Title: Uterine Skeletonization for Deep Infiltrative Endometriosis (DIE) Hysterectomy
Acronym: SKELETONDIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Baris KAYA, Associate Professor, Başakşehir Çam & Sakura City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-96317027-514.10-253796352; E-96317027-514.10-253796352 (Other: Basaksehir Cam ve Sakura City Hospital)
Record Dates: First submitted 2025-01-10; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Deep Infiltrating Endometriosis (DIE); Nerve Sparing Modified Radical Hysterectomy; Uterine Skeletonization
Keywords: Deep Infiltrating Endometriosis (DIE); Nerve sparing modified radical hysterectomy; Uterine skeletonization

STUDY DESIGN:
Intervention Model Description: Retrospective analysis of the prospectively collected data of the surgical technique, intraoperative and postoperative clinical outcomes and complications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- "Evaluation of Uterine Skeletonization-Based Nerve-Sparing Modified Radical Hysterectomy in Deep Inf (Other): Data on patients' demographics, preoperative treatments, imaging findings (ultrasound, CT, MRI), and surgical details (duration, type, complications) will be collected. Postoperative complications and pathological results of excised specimens will also be evaluated.
  Interventions: Procedure: Clinical Outcomes and Surgical Insights from Nerve-Sparing Hysterectomy with Uterine Skeletonization for Deep Infiltrative Endometriosis

INTERVENTIONS:
Procedure: Clinical Outcomes and Surgical Insights from Nerve-Sparing Hysterectomy with Uterine Skeletonization for Deep Infiltrative Endometriosis — In this retrospective study, the patents whom underwent nerve sparing modified radical hysterectomy for deeply infiltrating endometriosis with uterine skeletonization technique will be reviewed. The uterine skeletonization technique was developed by the princible investigator (BK) for DIE modified radical hsyterectomy and performed systematically in Basaksehir Cam ve Sakura City Hospital. The detailed surgical steps, surgical data such as operation duration, surgical type (e.g., hysterectomy + salpingo-oophorectomy, excision of parametrial, rectovaginal, or vaginal nodules, and bowel resections), and intraoperative complications (organ injuries, blood transfusions, conversion to open surgery) will be recorded. Early and late postoperative complications (fever, deep vein thrombosis, sepsis, pelvic abscess, genitourinary fistulas, anastomotic leaks, reoperation, vaginal cuff bleeding or abscess, and bladder dysfunction) will also be evaluated.

SUMMARY:
Endometriosis is characterized by the presence of endometrial glands and stroma outside the uterine cavity, accompanied by chronic inflammation. The most common locations of endometriosis are the ovaries, ovarian fossae, uterosacral ligaments, and the posterior cul-de-sac. Endometriosis lesions may be superficial, ovarian, or deeply infiltrative. Lesions that invade the rectovaginal space and/or the bowel are defined as deep infiltrative endometriosis (DIE). The invasive nature of these implants can lead to infertility, severe menstrual pain (dysmenorrhea), pain during intercourse (dyspareunia), and chronic pelvic pain. In cases of bowel involvement, symptoms such as constipation, painful defecation, and rectal bleeding may occur. When the urinary system is affected, patients may experience painful urination, hematuria, urinary dysfunction, and, in severe cases, renal loss due to ureteral obstruction.Treatment options vary depending on the severity and localization of the disease, the patient's desire for fertility, and their age. Treatment can include medical therapy, surgical therapy, or a combination of both. Surgical approaches to DIE can be conservative or definitive. Conservative surgery involves the removal of symptomatic endometriotic lesions without damaging surrounding structures. Definitive surgery typically includes hysterectomy with bilateral salpingo-oophorectomy and the excision of symptomatic lesions in other areas (e.g., peritoneum, bowel), often described as a radical hysterectomy. Here in this study, the hospital records of the patients who underwent modified radical nerve sapring hysterectomy for deeply infiltrating endometriosis by the gynecologist Baris Kaya,MD will be evaluated. The demographic and clinical characteristics of patients who underwent hysterectomy for endometriosis at our hospital's endometriosis clinic will be retrospectively analyzed. The diagnosis of these patients was already established through routine pelvic examination, transvaginal ultrasonography, and MRI at the endometriosis clinic of Basaksehir Cam ve Sakura City Hospital.

DETAILED DESCRIPTION:
The aim of this study is to contribute to the literature by evaluating the surgical features, intraoperative complications, and postoperative outcomes of patients undergoing nerve-sparing hysterectomy due to endometriosis. Steps of the modified radical hysterectomy for deeply infiltrating endometriosis with uterine skeletonization technique will be clearly stated, Data on patients' age, body mass index (BMI), known comorbidities, mode and number of deliveries, and previous surgeries will be collected, along with preoperative medical treatments. Visual analog scale (VAS) scores for dysmenorrhea, dyspareunia, dysuria, dyschezia, and chronic pelvic pain will be obtained from the HBYS system or patient files. Preoperative imaging findings, including ultrasonography, computed tomography (CT), and MRI, will be reviewed. Surgical data such as operation duration, surgical type (e.g., hysterectomy + salpingo-oophorectomy, excision of parametrial, rectovaginal, or vaginal nodules, and bowel resections), and intraoperative complications (organ injuries, blood transfusions, conversion to open surgery) will be recorded. ENZIAN scores according to the surgical findings will be stated. Early and late postoperative complications (fever, deep vein thrombosis, sepsis, pelvic abscess, genitourinary fistulas, anastomotic leaks, reoperation, vaginal cuff bleeding or abscess, and bladder dysfunction) will also be evaluated according to Clavien-Dindo Clasification. Pathological examination results of the excised specimens will be included.

ELIGIBILITY:
Inclusion Criteria:

Patients Aged 30-50

Patients with severe dysmenorrhea (VAS>7) dyspareunia (VAS>7), and /or diskhezia and/or chronic pelvic pain

Patients with deep infiltrating endometriosis who are unresponsive to medical treatment

Only patients who underwent nerve sparing hysterectomy by the principal investigator (BK)

Exclusion Criteria:

Patients under 30 or over 50 years of age. Patients who did not undergo nerve-sparing hysterectomy or salpingo-oophorectomy.

Patients with incomplete medical records or missing preoperative imaging data. Patients with a history of pelvic or abdominal malignancy. Patients with significant comorbidities such as advanced cardiovascular or respiratory diseases that may affect surgical outcomes.

Patients who responded positively to medical treatment and did not require surgical intervention.

Patients diagnosed with bowel, bladder, or rectovaginal fistulas unrelated to endometriosis.

Patients undergoing emergency surgeries unrelated to endometriosis. Patients unwilling to provide consent for their data to be used in the study.

-

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — endometriosis is a disease of biologically female gender
Enrollment: 75 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
1.Surgical features of the Modified Radical Hysterectomy for DIE with Uterine Sketelonization | From placing the laparoscopic trocars to the end of the surgery
  Surgical data such as detailed anatomical surgical steps of the surgery, surgery type (e.g., hysterectomy + salpingo-oophorectomy, excision of parametrial, rectovaginal, or vaginal nodules, and bowel resections)
Duration of operation | From placing the laparoscopic trocars to the end of the surgery
  Duration of the laparascopic deep infiltrating hysterectomy with uterine skeletonization will be stated which was recorded as minute.
Intraoperative complications | From placing the laparoscopic trocars to the end of the surgery
  Complications during surgery for deep infiltrating surgery such as bladder, ureter, bowel and nerve injuries will be reviewed.

SECONDARY OUTCOMES:
Postoperative complications | From enrollment to the end of treatment at 12 weeks
  Postoperative complications following surgery of the deep infiltrative endometriosis hysterectomy.
  Surgical site infections (SSI), urinary tract infections, or pelvic abscesses. Urogenital or rectovaginal fistulas following surgery. Vaginal Cuff Dehiscence, thromboembolic Events, Bladder or bowel dysfunction due to hypogastric and/or pelvic splanchnic nerve damages. These will also be stated as Clavien Dindo classification.

OTHER OUTCOMES:
Age of the patients | From enrollment to the end of treatment at 8 weeks
  Patients' age in years will be collected.
Patients' weight | From enrollment to the end of treatment at 8 weeks
  Patients' weight in kilograms will be collected.
Patients' height | From enrollment to the end of treatment at 8 weeks
  Patients' height will be stated as meters obtained from medical records.
Patients' BMI | From enrollment to the end of treatment at 8 weeks
  Body mass index of the patients will be calculated by weight (kg) and height (meter) will be combined to report BMI in kg/m^2
Patients' Medical History | From enrollment to the end of treatment at 8 weeks
  Known comorbidities, mode and number of deliveries, and previous surgeries will be collected, along with preoperative medical treatments from medical records .
Preoperative Imaging | From enrollment to the end of treatment at 8 weeks
  Preoperative imaging findings, including ultrasonography, computed tomography (CT), and Magnetic Resonance Imaging (MRI) reports, will be reviewed.
Visual analog scale (VAS) scores | From enrollment to the end of treatment at 12 weeks
  Visual analog scale (VAS) scores for dysmenorrhea, dyspareunia, dysuria, dyschezia, and chronic pelvic pain before and after the surgery will be obtained from the hospital records and patient files.

CONTACTS AND LOCATIONS:
Overall Officials: Baris Kaya, Associate Professor, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"Individual Participant Data (IPD) will not be shared due to privacy and confidentiality concerns. Additionally, resource limitations prevent proper preparation and documentation of IPD for external sharing."

REFERENCES:
- [Background] Nezhat C, Nguyen K, Ackroyd E, Roman RA, Rambhatla A, Nezhat A, Asiaii A. Nerve-Sparing Modified Radical Hysterectomy for Severe Endometriosis and Complex Pelvic Pathology. Cureus. 2020 Aug 19;12(8):e9882. doi: 10.7759/cureus.9882. PMID 32963921
- [Background] Rosati A, Pavone M, Campolo F, De Cicco Nardone A, Raimondo D, Serracchioli R, Scambia G, Ianieri MM. Surgical and functional impact of nerve-sparing radical hysterectomy for parametrial deep endometriosis: a single centre experience. Facts Views Vis Obgyn. 2022 Jun;14(2):121-127. doi: 10.52054/FVVO.14.2.016. PMID 35781108
- [Background] Muallem MZ, Diab Y, Sehouli J, Fujii S. Nerve-sparing radical hysterectomy: steps to standardize surgical technique. Int J Gynecol Cancer. 2019 Sep;29(7):1203-1208. doi: 10.1136/ijgc-2019-000410. Epub 2019 Jul 19. PMID 31326949
- [Background] Darwish B, Roman H. Nerve Sparing and Surgery for Deep Infiltrating Endometriosis: Pessimism of the Intellect or Optimism of the Will. Semin Reprod Med. 2017 Jan;35(1):72-80. doi: 10.1055/s-0036-1597305. Epub 2016 Dec 12. PMID 27951614